CLINICAL TRIAL: NCT03779997
Title: Development and Evaluation of Video-Based Directly Observed Therapy for Office-Based Treatment of Opioid Use Disorders With Buprenorphine
Brief Title: Trial of Adherence App for Buprenorphine Treatment (TAAB) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); emocha Mobile Health, Inc. (Other)
Responsible Party: Principal Investigator, Judith I. Tsui, Associate Professor of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005069; 4R44DA044053-02 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-06

CONDITIONS: Opioid-Related Disorders
Keywords: Buprenorphine; Directly Observed Therapy; mHealth; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Directly Observed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-based DOT Application (Experimental)
  Interventions: Behavioral: Video-based DOT Application
- Treatment as Usual (TAU) (No Intervention)

INTERVENTIONS:
Behavioral: Video-based DOT Application — Participants will be asked to record daily videos of themselves confirming daily ingestion of their buprenorphine. Clinical staff (i.e. physicians, nurses and medical assistants) of patients enrolled in the intervention group will be given training and the opportunity to review medication taking videos.
  Arms: Video-based DOT Application

SUMMARY:
The purpose of this study is to pilot test a smartphone application that allows video-based directly observed therapy for participants receiving buprenorphine treatment for opioid use disorder in office-based settings. This application may help participants take their medication more regularly so that they are successful in treatment. Participants will be randomly assigned to either using a smartphone application that allows them to take daily videos confirming their buprenorphine medication ingestion or they will continue with their care as usual (treatment-as-usual or TAU). The primary study outcome will be the percentage of weekly study urine drug tests that are negative for opiates between baseline and 12 weeks post-randomization. The secondary outcome will be engagement in treatment at week 12.

DETAILED DESCRIPTION:
The objective of this study is to compare an innovative mobile health (mHealth) platform to support participants being treated for opioid use disorder (OUD) with buprenorphine to treatment-as-usual (TAU). The application will provide video-based directly observed therapy (VDOT) which may result in better health outcomes for participants and less public health risk for diversion. This study is a randomized controlled trial with two arms: TAU and mHealth intervention. Randomization to the two study arms will be completed using computer randomization procedures. Participants in the intervention group will learn how to use the mHealth application on their personal smartphones or tablets. If a participant does not have access to a personal device or prefers to not use a personal device then a study-provided smartphone will be offered for the duration of the study. Intervention participants are asked to record one daily video of themselves taking buprenorphine. Buprenorphine clinical staff (i.e., physicians, nurses and medical assistants) of patients enrolled in the intervention group will be trained and have the opportunity to review the videos. Adherence for the intervention group will be measured through participation in VDOT, namely the percentage of daily medication doses that are observed through submitted videos. The TAU group will not be given access to the intervention and therefore will not have the opportunity to be exposed to the intervention.

All participants will follow the same visit schedule. Interviews will occur at baseline (Week 0) and the final visit (Week 12) to assess current and prior substance use, treatment history, medication adherence, drug diversion, general physical and mental health and treatment satisfaction. A point of care urine drug test will also be administered which will assess for opiates and other substances. In between the baseline and final visits, participants will meet with research staff weekly to conduct a urine drug test and assess self-reported adherence to buprenorphine. Research staff will review the electronic medical record at baseline and week 12 to assess engagement in treatment. Additionally, at 24 weeks post-enrollment the research staff will complete a review of the electronic medical record and record engagement in clinic treatment, changes in buprenorphine treatment during the study period and the results of any clinical urine drug testing.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Receiving buprenorphine treatment at an office-based buprenorphine program for ≤4 weeks
* Willing to be randomized to either VDOT or TAU

Exclusion Criteria:

* Unable or unwilling to use smart phone
* Cognitive impairment resulting in inability to provide informed consent
* Researcher's discretion that participant will not be appropriate for participation in the study (e.g. participant is planning on moving away, is knowledgeable of future incarceration during the study, or has behavioral issues that may pose safety concerns for clinic and research staff)
* Inability to read and understand English as needed for following app instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith I. Tsui, MD, MPH, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Boston University, Boston, Massachusetts
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schramm ZA, Leroux BG, Radick AC, Ventura AS, Klein JW, Samet JH, Saxon AJ, Kim TW, Tsui JI. Video directly observed therapy intervention using a mobile health application among opioid use disorder patients receiving office-based buprenorphine treatment: protocol for a pilot randomized controlled trial. Addict Sci Clin Pract. 2020 Jul 31;15(1):30. doi: 10.1186/s13722-020-00203-9. PMID 32736660
- [Result] Tsui JI, Leroux BG, Radick AC, Schramm ZA, Blalock K, Labelle C, Heerema M, Klein JW, Merrill JO, Saxon AJ, Samet JH, Kim TW. Video directly observed therapy for patients receiving office-based buprenorphine - A pilot randomized controlled trial. Drug Alcohol Depend. 2021 Oct 1;227:108917. doi: 10.1016/j.drugalcdep.2021.108917. Epub 2021 Jul 28. PMID 34399136
- [Derived] Radick AC, James J, Leroux BG, Kim TW, Saxon AJ, Samet JH, Tsui JI. Use of Video Directly Observed Therapy and Characteristics Associated With Use Among Patients Treated With Buprenorphine in an Office-based Setting. J Addict Med. 2023 May-Jun 01;17(3):300-304. doi: 10.1097/ADM.0000000000001103. Epub 2022 Oct 25. PMID 37267172

RESULTS

PARTICIPANT FLOW:
Groups:
- Video-based DOT Application: Video-based directly observed therapy (DOT) Application: Participants will be asked to record daily videos of themselves confirming daily ingestion of their buprenorphine. Clinical staff (i.e. physicians, nurses and medical assistants) of patients enrolled in the intervention group will be given training and the opportunity to review medication taking videos.
- Treatment as Usual (TAU): Treatment-as-usual administered at office-based buprenorphine treatment clinics.
Period: Overall Study
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Started | 39 | 39
Completed at Least One Visit | 39 | 39
Completed | 39 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual (TAU): Office-based buprenorphine treatment
- Total: Total of all reporting groups
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.9) | 40.7 (12.0) | 41.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 29 | 29 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 6 | 2 | 8
  White | 23 | 25 | 48
  More than one race | 4 | 9 | 13
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78
Study Site [Count of Participants; unit: Participants] — Site of enrollment
  Participants
    Seattle | 19 | 19 | 38
    Boston | 20 | 20 | 40
Education [Count of Participants; unit: Participants] — Self-reported participant education level
  Participants
    Less than a high school diploma | 7 | 6 | 13
    High school diploma/GED | 13 | 20 | 33
    Some post-high school | 9 | 9 | 18
    College degree | 9 | 4 | 13
    Postgraduate | 1 | 0 | 1
Prior Buprenorphine Treatment [Count of Participants; unit: Participants] — Self-report at baseline of receiving prior buprenorphine treatment prescribed by a doctor (No/Yes).
  Participants
    No | 15 | 19 | 34
    Yes | 24 | 20 | 44
Homelessness [Count of Participants; unit: Participants] — Self-reported baseline homelessness within the past 3 months.
  Participants
    Not homeless | 24 | 23 | 47
    Homeless | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage Opioid Negative Urine Tests
Description: Percentage of weekly study urine drug tests that are negative for opioids, missing assumed to be positive.
Time Frame: Baseline to 12 weeks post-randomization
Measure: Count of Units; unit: urine drug tests
Units Other Than Participants: urine drug tests
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 39
Number analyzed (urine drug tests) | 468 | 468
urine drug tests | 234 | 299
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: no difference in the percentage of urine drug tests (UDT) negative for opioids between the two treatment arms.Treatment-as-usual (TAU) is the reference group; Test type: Superiority; p = 0.07, Log-linear GEE regression — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.60 to 1.02], Standard Deviation 0.10

2. Secondary Outcome: Percentage of Participants Engaged in Treatment at Week 12
Description: The percentage of participants with an active script for buprenorphine at week 12 (engaged in treatment), measured by electronic health record (EHR) review.
Time Frame: Week 12 post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 39
Participants | 27 | 32
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: no difference between treatment arms in the percentage of patients engaged in treatment at week 12. TAU is the reference group; Test type: Superiority; p = 0.20, Poisson regression with robust SEs — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.65 to 1.10], Standard Deviation 0.11

3. Other Pre Specified Outcome: Percentage of Participants Engaged in Treatment at Week 24
Description: The percentage of participants engaged in treatment at 24 weeks post-randomization, measured by EHR review.
Time Frame: Week 24 post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 39
Participants | 16 | 22
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms in the percentage of participants engaged in treatment at week 24 post-randomization. TAU is the reference group; Test type: Superiority; p = 0.18, Poisson regression with robust SEs — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.45 to 1.16], Standard Deviation 0.17

4. Other Pre Specified Outcome: Consecutive Weeks Opioid Negative Urine Tests
Description: The number of consecutive weeks with urine drug test negative for opioids.
Time Frame: Baseline to 12 weeks post-randomization
Measure: Mean (Standard Deviation); unit: weeks
Units Other Than Participants: Weeks
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 39
Number analyzed (Weeks) | 12 | 12
weeks | 4.8 (4.2) | 5.7 (3.7)
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms on the number of consecutive weeks with UDT negative for opioids; Test type: Superiority; p = 0.31, t-test, 2 sided — 0.05 a priori threshold for statistical significance; Median Difference (Final Values) = 0.9, 95% CI 2-sided [-0.9 to 2.7], Standard Deviation 0.45 — TAU is the reference group

5. Other Pre Specified Outcome: Number of Participants With Self-report of Opioid Use
Description: Self-reported use of illicit opioids in past 30 days at week 12.
Time Frame: Week 12 post-randomization
Population: There were 15 missing survey responses among the video DOT application arm and 9 missing from the TAU arm, these participants were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 30
Participants | 4 | 7
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms in the number of participants who self-reported illicit opioid use at week 12; Test type: Superiority; p = 0.57, Poisson regression with robust SEs — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 0.71, 95% CI 2-sided [0.23 to 2.26], Standard Deviation 0.41 — TAU is the reference group

6. Other Pre Specified Outcome: Buprenorphine Adherence Self-Report
Description: Mean number of days adherent to buprenorphine by self-report over the 12-week study period, using a 7-day timeline-follow-back (TLFB) survey procedure each week. Days with missing data were excluded from analysis.
Time Frame: Baseline to 12 weeks post-randomization
Population: Missing days are excluded from analysis.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: Days
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 39
Number analyzed (Days) | 281 | 378
days | 5.99 (2.18) | 5.93 (2.10)
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms in the mean number of days adherent to buprenorphine by self-report; Test type: Superiority; p = 0.88, GEE Poisson regression — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.89 to 1.15], Standard Deviation 0.066 — TAU is the reference group

7. Other Pre Specified Outcome: Treatment Discharge
Description: Time to discharge from treatment, measured by EHR review.
Time Frame: Baseline to 24 weeks post-randomization
Population: Data was not avaiable on video-based DOT application participants. Therefore, data analysis is not possible.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 0 | 4
Days |  | NA (NA) — Data collected on only 4 participants.

8. Other Pre Specified Outcome: Buprenorphine Non-use: One or More UDT Negative for Buprenorphine
Description: Having one or more study urine drug tests negative for buprenorphine
Time Frame: Baseline to 12 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 39 | 39
Participants | 7 | 6
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms in number of participants who had one or more urine drug tests negative for buprenorphine; Test type: Superiority; p = 0.77, Poisson regression with robust SEs — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.42 to 3.24], Standard Deviation 0.60 — TAU is the reference group

9. Other Pre Specified Outcome: UDT Positive for Stimulants at Week 12
Description: Number of participants having a study urine drug test positive for stimulants (cocaine, amphetamines or methamphetamines).
Time Frame: Week 12 post-randomization
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 30
Participants | 7 | 13
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms in number of participants who tested positive for stimulants at week 12; Test type: Superiority; p = 0.30, Poisson regression with robust SEs — 0.05 a priori threshold for statistical significance; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.32 to 1.43], Standard Deviation 0.26 — TAU is the reference group

10. Other Pre Specified Outcome: Treatment Satisfaction
Description: Likert scale survey question of participant's satisfaction with clinic's treatment of opioid use disorder (OUD); on a scale of 1-5, with 1 being very dissatisfied and 5 being very satisfied.
Time Frame: Week 12 post-randomization
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
Number analyzed (Participants) | 24 | 30
score on a scale | 4.6 (0.6) | 4.6 (0.5)
Statistical Analysis 1: Comparison: Video-based DOT Application vs Treatment as Usual (TAU); Null hypothesis: No difference between arms in mean treatment satisfaction scores; Test type: Superiority; p = 0.91, t-test, 2 sided — 0.05 a priori threshold for statistical significance; Median Difference (Final Values) = 0.02, 95% CI 2-sided [-0.29 to 0.32], Standard Deviation 0.07 — TAU is the reference group

ADVERSE EVENTS:
Time Frame: Up to 24 weeks.
Arm/Group | Video-based DOT Application | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 1/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 9/39 | 3/39
Other Adverse Events (participants affected / at risk) | 3/39 | 1/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video-based DOT Application (N=39) | Treatment as Usual (TAU) (N=39)
In-patient hospitalization (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
In-patient hospitalization (Psychiatric disorders) | 4 (4) | 2 (2)
In-patient hospitalization (Infections and infestations) | 1 (1) | 0 (0)
In-patient hospitalization (Cardiac disorders) | 1 (1) | 1 (1)
In-patient hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
In-patient hospitalization (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Video-based DOT Application (N=39) | Treatment as Usual (TAU) (N=39)
Nausea from medicine (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain - lower extremities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generall Illness (General disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the study included a small sample size and limited power for detecting small but clinically meaningful differences in outcomes. The study did not provide participants with incentives for using the intervention, which may have resulted in low rates of use. Limited provider and clinic staff involvement in the intervention is another limitation that may have affected the uptake of video DOT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT03779997/Prot_SAP_000.pdf